CLINICAL TRIAL: NCT06424158
Title: The Impact of Massage Therapy on Post-Surgical Pain, Anxiety, Quality of Life, and Opioid Analgesia Exposure on Children After Thoracic or Lumbar Surgery
Brief Title: Massage Therapy After Thoracic or Lumbar Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cook Children's Health Care System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020-088
Record Dates: First submitted 2024-04-05; First posted 2024-05-22 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Scoliosis; Adolescence; Adolescent Idiopathic Scoliosis, Thoracic Region; Adolescent Idiopathic Scoliosis, Lumbar Region
Keywords: Spinal Fusion; Massage Therapy; Pain Management; Scoliosis
MeSH Terms: conditions — Scoliosis; Agnosia | interventions — Massage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Massage Therapy Group (Experimental): Participants in the massage therapy group are treated by a certified pediatric massage therapist for at least two 30- minute massage therapy sessions performed on postoperative days two and four or five. Participants will continue to receive standard of care, including any pain medications as needed.
  Interventions: Other: Massage Therapy
- Control Group (No Intervention): Participants in control group will continue to receive the normal standard of care as usual for their recovery and will be monitored by hospital staff in obtaining the same data points recorded clinically for post-op days 2 and 4/5; however, no therapeutic intervention will occur.

INTERVENTIONS:
Other: Massage Therapy — Massage therapy (MT) has been proven as an alternative non-opioid pain management intervention, particularly towards reducing pain, diminishing depression, improving immune function, and increasing alertness in the adult population. MT raises the temperature of local tissues, dilates capillaries, accelerates the circulation of blood and lymph, promotes the absorption of local tissue metabolism and mass inflammation, improves the nutritional supply of surrounding muscle groups, promotes their growth and development, and relieves pain.
  Arms: Massage Therapy Group

SUMMARY:
The purpose of this research is to look at the effect of massage therapy on the pain, anxiety, and quality of life that pediatric patients have after undergoing spinal fusion surgery. This is a single-site, prospective, randomized, interventional study design that will involve post-thoracic and post-lumbar spinal fusion surgeries of pediatric patients from 7 to 19 years of age that present to Cook Children's Medical Center in Fort Worth, Texas. These patients will be identified prior to their scheduled spinal fusion surgery and recruited to enroll in the study. The planned spinal fusion surgeries are not considered part of this research project, but rather considered standard of care and would occur whether the patient is enrolled in this project or not. Enrolled participants will be followed during their inpatient stay and through their subsequent follow-up visits at weeks 2, 6, and 12. Participants will be randomly assigned to either a massage therapy group or a group that receives the standard (normal) care for recovery after surgery. The final study involvement will occur at week 16 (post-hospital discharge) where a study team member will administer a quality of life (PedsQL) questionnaire via phone or mail with the subject. Data will be collected after study related procedures are completed.

DETAILED DESCRIPTION:
There has been an increasing amount of spinal fusion surgeries in the United States. These patients struggle with anxiety and stress before surgery, and experience significant hardship during postoperative recovery including management of opioid related side effects, effective pain control, delay in mobilization, and prolonged length of stay. A growing body of research, however, has shown massage therapy (MT) as an effective alternative to conventional treatments. MT raises the temperature of local tissues, dilates capillaries, accelerates the circulation of blood and lymph, promotes the absorption of local tissue metabolism and mass inflammation, improves the nutritional supply of surrounding muscle groups, promotes their growth and development, and relieves pain.

The aim of this present study is to assess the effect of MT on perceived post-surgical pain, anxiety, and quality of life experienced by pediatric patients who have undergone thoracic and lumbar spinal fusion.

Potential participants will be identified prior to their scheduled spinal fusion surgery and recruited to enroll in the study. The planned spinal fusion surgeries are not considered part of this research project, but rather considered standard of care and would occur whether the patient is enrolled in this project or not. After surgery, another review of inclusion and exclusion criteria will be done to determine the subject's continued eligibility for participation. If criteria are met, the child participant will be randomized into one of two study groups, 1) Massage Therapy Group or 2) A Control Group for their post-surgery recovery plan. Enrolled participants will be followed during their inpatient stay and through their subsequent follow-up visits at weeks 2, 6, and 12. The final study involvement will occur at week 16 (post-hospital discharge) where a study team member will administer a quality of life questionnaire via phone or mail with the subject.

All participants whom are randomized into the massage therapy group are treated by a certified pediatric massage therapist. At least two 30- minute massage therapy sessions are performed on postoperative days two and four or five. Either post-operative day 4 or 5 can be selected as a second in-patient massage therapy session as long as the session occurs Monday through Friday, as the massage therapy service is not offered during the weekend hours of Saturday or Sunday. If the participant's length of stay is six days or longer, the participant continues to receive treatment every other day for the duration of hospitalization. Each individual patient is treated according to what their needs are, which means one participant may prefer neck and shoulder massage and another may prefer legs and feet. The participant remains in a position of comfort which for spinal fusion patients is generally in the supine, sitting, or side laying position. A combination of therapies including myofascial release, compression, and Swedish massage will be employed. Light and medium touch are applied but never deep tissue. While scar mobilization is a desired outcome postoperatively, this is not an immediate goal. The incision site remains clean and covered without any manipulation. Rehabilitation goals are to maximize mobility and flexibility of surrounding structures but is only addressed by the physical therapy team. Massage therapy does not involve any form of stretching or range of motion techniques. The study team will obtain vital data (Blood Pressure, Heart Rate, and O2 stats) along with VAS pain scale and anxiety rating scale measures before and after every session from the patient's medical records.

For those participants randomized into the control group, they will continue to receive the normal standard of care as usual for their recovery and will be monitored by hospital staff in obtaining the same data points (e.g., BP values, HR value, O2 levels) recorded clinically for post-op days 2 and 4/5; as the investigators are collecting in the massage group; however, no therapeutic intervention will occur. If the participant's length of stay is greater than five days the study staff will continue to record these values every other day for the duration of hospitalization. Study staff will retrieve these data variables via the patient's electronic medical record and enter data into the study database. A study member will visit with the subject on day 2, day 4/5 (and every other day if length of stay is greater than five days) to collect anxiety and pain scores measurements.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo their first thoracic or lumbar spinal fusion surgery
* Able to participate and perform in a massage therapy as a recovery option
* Participant needs to be verbal
* Ability to understand study procedures and to comply with them for the entire length of the study

Exclusion Criteria:

* Prospective patients scheduled to undergo any spinal fusion other than a thoracic or lumbar spinal fusion surgery.
* Prospective patients scheduled to undergo a second or multiple thoracic or lumbar spinal fusion surgery
* Previous cardiac surgery
* Chronic pain syndromes
* Chronic opioid usage
* History of psychosis
* Prolonged bleeding
* Intubation greater than 24 hours
* Illicit/recreation drug use
* Paralysis diagnosis
* History of chronic pain requiring medical intervention
* Neuromuscular scoliosis diagnosis
* Cerebral palsy diagnosis
* Developmental delay characteristics

Ages: 7 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-02-17 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Pediatric Pain - Short Form (Neuro-QOL™) | Post-op day 2, day 4/5, week 2, week 6, and week 12
  A pain scale with 10 items. Responses range from "Never" (1) to "Almost Always" (5) with the minimum score being 10 and the maximum score being 50. Higher scores indicate worse outcome.
Visual Analogue Scale (VAS) Pain Rating Scale | Post-op day 2, day 4/5, week 2, week 6, and week 12
  A pain scale with one question asking patients to choose a number from 0 to 10 that best describes their pain from "No Pain" (0) to "Unbearable Pain" (10) with the minimum score being 0 and the maximum being 10. Higher scores indicate worse outcome.
Wong-Baker FACES® Pain Rating Scale | Post-op day 2, day 4/5, week 2, week 6, and week 12
  A pain scale with one question asking patients to choose a number from 0 to 5 that best describes their pain from "No Hurt" (0) to "Hurts Worst" (10) with the minimum score being 1 and the maximum score being 5. Higher scores indicate worse outcome.

SECONDARY OUTCOMES:
Pediatric Anxiety (PROMIS®) | Post-op day 2, day 4/5, week 2, week 6, and week 12
  An anxiety measure with 14 statements. Responses range from "Never" (1) to "Almost Always" (5). with the minimum score being 14 and the maximum being 70. Higher scores indicate worse outcome.
Anxiety Thermometer | Post-op day 2, day 4/5, week 2, week 6, and week 12
  An anxiety scale with one question asking patients to choose a number between 1 "Calm and content" and 10 "Extremely anxious, unable to function" that best describes their level of anxiety. The minimum score is 1 and the maximum score is 10. Higher scores indicate worse outcome.
Blood pressure | Post-op day 2, day 4/5, week 2, week 6, and week 12
  Measured as systolic blood pressure over diastolic blood pressure in units of millimeters of mercury (mmHg)
Heart Rate | Post-op day 2, day 4/5, week 2, week 6, and week 12
  Measured as beats per minute
Respiratory Rate | Post-op day 2, day 4/5, week 2, week 6, and week 12
  Oxygen saturation (%) measured before and after the participant's designated intervention
Pediatric Quality of Life Inventory (PedsQL™) | Baseline, and weeks 6, 12 and 16 post-op
  A quality of life scale with 15 questions. Responses range from "Never" (1) to "Almost Always" (5) with the minimum score being 15 and the maximum being 75. Higher scores indicate worse outcome.
Use of opioid analgesics post-surgery | Immediately after surgery, daily for up to 7 days after surgery, week 2, week 6, and week 12
  Count of opioid doses administered

OTHER OUTCOMES:
Scoliosis Patient Questionnaire (SRS-30) | Baseline and 12-week post-op
  A questionnaire with 30 questions related to health-related quality of life. Each question is scored on 1-5 scale with the minimum value being 30 and the maximum 150. Higher scores indicate worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Meredith Brooks, MD, Principal Investigator — Cook Children's Health Care System
Locations (1):
- Cook Children's Medical Center, Fort Worth, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] American Massage Therapy Association. Massage Therapy Industry Fact Sheet. (2019). American Massage Therapy Association website. https://www.amtamassage.org/globalassets/documents/src/2019-pdf.pdf. Published 2019. Accessed June 22, 2020.
- [Background] Bauer BA, Cutshall SM, Wentworth LJ, Engen D, Messner PK, Wood CM, Brekke KM, Kelly RF, Sundt TM 3rd. Effect of massage therapy on pain, anxiety, and tension after cardiac surgery: a randomized study. Complement Ther Clin Pract. 2010 May;16(2):70-5. doi: 10.1016/j.ctcp.2009.06.012. Epub 2009 Jul 14. PMID 20347836
- [Background] Beider S, Moyer CA. Randomized controlled trials of pediatric massage: a review. Evid Based Complement Alternat Med. 2007 Mar;4(1):23-34. doi: 10.1093/ecam/nel068. Epub 2006 Nov 3. PMID 17342238
- [Background] Braun LA, Stanguts C, Casanelia L, Spitzer O, Paul E, Vardaxis NJ, Rosenfeldt F. Massage therapy for cardiac surgery patients--a randomized trial. J Thorac Cardiovasc Surg. 2012 Dec;144(6):1453-9, 1459.e1. doi: 10.1016/j.jtcvs.2012.04.027. Epub 2012 Sep 7. PMID 22964355
- [Background] Blanco JS, Perlman SL, Cha HS, Delpizzo K. Multimodal pain management after spinal surgery for adolescent idiopathic scoliosis. Orthopedics. 2013 Feb;36(2 Suppl):33-5. doi: 10.3928/01477447-20130122-55. PMID 23379574
- [Background] Connelly M, Fulmer RD, Prohaska J, Anson L, Dryer L, Thomas V, Ariagno JE, Price N, Schwend R. Predictors of postoperative pain trajectories in adolescent idiopathic scoliosis. Spine (Phila Pa 1976). 2014 Feb 1;39(3):E174-81. doi: 10.1097/BRS.0000000000000099. PMID 24173016
- [Background] Erdogmus CB, Resch KL, Sabitzer R, Muller H, Nuhr M, Schoggl A, Posch M, Osterode W, Ungersbock K, Ebenbichler GR. Physiotherapy-based rehabilitation following disc herniation operation: results of a randomized clinical trial. Spine (Phila Pa 1976). 2007 Sep 1;32(19):2041-9. doi: 10.1097/BRS.0b013e318145a386. PMID 17762803
- [Background] Falkensteiner M, Mantovan F, Muller I, Them C. The use of massage therapy for reducing pain, anxiety, and depression in oncological palliative care patients: a narrative review of the literature. ISRN Nurs. 2011;2011:929868. doi: 10.5402/2011/929868. Epub 2011 Aug 23. PMID 22007330
- [Background] Field TM, Quintino O, Hernandez-Reif M, Koslovsky G. Adolescents with attention deficit hyperactivity disorder benefit from massage therapy. Adolescence. 1998 Spring;33(129):103-8. PMID 9583664
- [Background] Field T, Grizzle N, Scafidi F, Schanberg S. Massage and relaxation therapies' effects on depressed adolescent mothers. Adolescence. 1996 Winter;31(124):903-11. PMID 8970662
- [Background] Field T, Morrow C, Valdeon C, Larson S, Kuhn C, Schanberg S. Massage reduces anxiety in child and adolescent psychiatric patients. J Am Acad Child Adolesc Psychiatry. 1992 Jan;31(1):125-31. doi: 10.1097/00004583-199201000-00019. PMID 1537763
- [Background] Gan TJ, Habib AS, Miller TE, White W, Apfelbaum JL. Incidence, patient satisfaction, and perceptions of post-surgical pain: results from a US national survey. Curr Med Res Opin. 2014 Jan;30(1):149-60. doi: 10.1185/03007995.2013.860019. Epub 2013 Nov 15. PMID 24237004
- [Background] Jadhav MP, Jadhav PM, Shelke P, Sharma Y, Nadkar M. Assessment of use of complementary alternative medicine and its impact on quality of life in the patients attending rheumatology clinic, in a tertiary care centre in India. Indian J Med Sci. 2011 Feb;65(2):50-7. PMID 23196313
- [Background] Kain ZN. Postoperative maladaptive behavioral changes in children: incidence, risks factors and interventions. Acta Anaesthesiol Belg. 2000;51(4):217-26. No abstract available. PMID 11129622
- [Background] Kain ZN, Mayes LC, O'Connor TZ, Cicchetti DV. Preoperative anxiety in children. Predictors and outcomes. Arch Pediatr Adolesc Med. 1996 Dec;150(12):1238-45. doi: 10.1001/archpedi.1996.02170370016002. PMID 8953995
- [Background] Martin CT, Pugely AJ, Gao Y, Mendoza-Lattes SA, Ilgenfritz RM, Callaghan JJ, Weinstein SL. Increasing hospital charges for adolescent idiopathic scoliosis in the United States. Spine (Phila Pa 1976). 2014 Sep 15;39(20):1676-82. doi: 10.1097/BRS.0000000000000501. PMID 24983937
- [Background] Mathews L. Pain in children: neglected, unaddressed and mismanaged. Indian J Palliat Care. 2011 Jan;17(Suppl):S70-3. doi: 10.4103/0973-1075.76247. PMID 21811376
- [Background] McGregor AH, Dore CJ, Morris TP, Morris S, Jamrozik K. Function after spinal treatment, exercise and rehabilitation (FASTER): improving the functional outcome of spinal surgery. BMC Musculoskelet Disord. 2010 Jan 26;11:17. doi: 10.1186/1471-2474-11-17. PMID 20102625
- [Background] Muhly WT, Sankar WN, Ryan K, Norton A, Maxwell LG, DiMaggio T, Farrell S, Hughes R, Gornitzky A, Keren R, McCloskey JJ, Flynn JM. Rapid Recovery Pathway After Spinal Fusion for Idiopathic Scoliosis. Pediatrics. 2016 Apr;137(4):e20151568. doi: 10.1542/peds.2015-1568. Epub 2016 Mar 23. PMID 27009035
- [Background] Noshchenko A, Hoffecker L, Lindley EM, Burger EL, Cain CM, Patel VV, Bradford AP. Predictors of spine deformity progression in adolescent idiopathic scoliosis: A systematic review with meta-analysis. World J Orthop. 2015 Aug 18;6(7):537-58. doi: 10.5312/wjo.v6.i7.537. eCollection 2015 Aug 18. PMID 26301183
- [Background] Rumalla K, Yarbrough CK, Pugely AJ, Koester L, Dorward IG. Spinal fusion for pediatric neuromuscular scoliosis: national trends, complications, and in-hospital outcomes. J Neurosurg Spine. 2016 Oct;25(4):500-508. doi: 10.3171/2016.2.SPINE151377. Epub 2016 May 20. PMID 27203810
- [Background] Smith SL, Lux R, Haley S, Slater H, Beachy J, Moyer-Mileur LJ. The effect of massage on heart rate variability in preterm infants. J Perinatol. 2013 Jan;33(1):59-64. doi: 10.1038/jp.2012.47. Epub 2012 Apr 26. PMID 22538325
- [Background] Staveski SL, Boulanger K, Erman L, Lin L, Almgren C, Journel C, Roth SJ, Golianu B. The Impact of Massage and Reading on Children's Pain and Anxiety After Cardiovascular Surgery: A Pilot Study. Pediatr Crit Care Med. 2018 Aug;19(8):725-732. doi: 10.1097/PCC.0000000000001615. PMID 29912070
- [Background] Theologis AA, Sing DC, Chekeni F, Diab M. National Trends in the Surgical Management of Adolescent Idiopathic Scoliosis: Analysis of a National Estimate of 60,108 Children From the National Inpatient Sample Over a 13-Year Time Period in the United States. Spine Deform. 2017 Jan;5(1):56-65. doi: 10.1016/j.jspd.2016.09.001. PMID 28038695
- [Background] Yang S, Werner BC. Risk Factors for Prolonged Postoperative Opioid Use After Spinal Fusion for Adolescent Idiopathic Scoliosis. J Pediatr Orthop. 2019 Nov/Dec;39(10):500-504. doi: 10.1097/BPO.0000000000001139. PMID 31599858